CLINICAL TRIAL: NCT05161455
Title: Extraction and Socket Preservation Before Implant Placement Using Freezed Dried Allograft (FDBA) and Platelet-Rich Fibrin in Smokers. A Single Blinded Randomized Controlled Clinical Trial
Brief Title: Extraction and Socket Preservation Before Implant Placement Using Freezed Dried Allograft (FDBA) and Platelet-Rich Fibrin in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, yasser fahad alrayyes, Doctor, PHD student, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-21-5999
Record Dates: First submitted 2021-11-12; First posted 2021-12-17 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: A-PRF

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A-PRF (Experimental)
  Interventions: Biological: platelet rich fibrin
- A-PRF+ allograft bone (Experimental)
  Interventions: Biological: platelet rich fibrin
- allograft bone+crosslinked collagen membrane (Active Comparator)
  Interventions: Biological: platelet rich fibrin
- collagen plug (Sham Comparator)
  Interventions: Biological: platelet rich fibrin

INTERVENTIONS:
Biological: platelet rich fibrin — we would like to measure the effect of PRF on soft and hard tissue healing

SUMMARY:
the investigators aim from this study to evaluate platelet rich fibrin potential to heal the periodontal tissue and to form new native bone in smokers that require socket augmentation following dental extraction and before implant placement.

Materials and Methods: 18 adult smoker patients with 40 extracted sockets were recruited for this study, and the extracted sockets were distributed into four different groups as follows; Group 1- A-PRF alone, Group 2- Factors-enriched bone graft matrix (commonly known as sticky bone) using autologous fibrin glue combined with an FDBA with CGF-Enriched Fibrin Membrane to covered it, Group 3- an FDBA with a crosslinked collagen membrane and Group 4-Resorbable collagen plug (RCP) alone serving as a negative control group.

The patients were randomly grouped into a previously mentioned group, and the socket dimensions were measured four times, immediately after the extraction (0 days), after 10, 21, and 28 days to assess epithelial layer healing.

After six months and before placing the implant fixture, both soft and hard tissue samples will be harvested to be evaluated and compared histologically, also standardized CBCT will be taken before and after extraction to evaluate the amount of mineral content and vital bone formation radiographically.

ELIGIBILITY:
* Inclusion Criteria:

  * Current smokers
  * have at least one tooth indicated for extraction due to extensive decay, tooth fracture or failed root canal treatment.
  * 21 years of age or older.
  * give a written consent to participate in the trial.
  * have the desire to have an implant restoration for at least one non-restorable tooth
  * indicated for socket preservation procedures and generally healthy with no systematic disease
* Exclusion Criteria:

  * subjects who unable to undergo oral surgery procedures due to a medical condition.
  * women who are pregnant or nursing a child.
  * subjects with dental infection of bone, active periodontal disease and ankylosed teeth.
  * Subjects with following systemic diseases and conditions: Chemotherapy or radiation for the treatment of cancer and arthritis, seriously impaired cardiovascular or pulmonary function, uncontrolled diabetes, auto-immune compromised diseases, kidney or liver disease and history of severe, multiple allergies.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
soft tissue healing and migration. | 28 days
  In all groups, the buccolingual and mesiodistal dimensions at the osseous crest of the extraction socket will be measured at the midpoints immediately after extraction with a University of Michigan O Probe with Williams marking (Hu-Friedy® Mfg Chicago, IL, USA) at 0, 10, 21, and 28 days.
bone height after ridge preservation. | 6 months
  two different measurements shall be taken at baseline and after 6 months using Cone-beam computed tomography to asess vertical resorption measured by mean difference in length of socket.
bone width after ridge preservation. | 6 months
  two different measurements shall be taken at baseline and after 6 months using Cone-beam computed tomography to asess the mean width ridge difference between outer border of buccal and lingual cortical plate at Socket depth at 1, 3,5 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided